CLINICAL TRIAL: NCT06089499
Title: The PACED Study: A Randomized Controlled Pilot Study of Palliative Care Education Compared to Usual Care on Health Literacy and Quality of Life Among Older Adults With Chronic Obstructive Pulmonary Disease
Brief Title: Palliative Care Health Literacy Education and QOL Compared to Usual Care
Acronym: PACED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Kelly Counts, Principal Investigator, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB#2096893-AA
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: COPD
Keywords: Health Literacy QOL Palliative Care COPD; Emergency Medicine Older Adults
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Recruitment will take place for 30 days, and the study duration will be 30 days from the time of enrollment. A 1:1 randomization will be used to assign participants to the treatment or control group. The goal of 15 participants in each arm of the pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Get Palliative Care: four educational learning module videos (Experimental): Get Palliative Care educational learning module videos available online in the public domain. A Webinar: How to Manage Shortness of Breath and Improve Your Quality of Life (2019) presented by Tara Liberman, DO reviews how to live with COPD, where and when palliative care can be implemented, what alternatives to treatment may look like, and final provides a summary of the benefits of palliative care. Each learning module is approximately five to seven minutes in length. The four learning modules are accessible at https://youtu.be/__phRXS4jZs?si=TivFch6cFE6roXDZ. After completing the weekly learning module, the participant will log their viewing in REDCap via a link provided to the participant by the email provided at the time of enrollment.
  Interventions: Behavioral: Get Palliative Care: four educational learning module videos
- Usual Care (No Intervention): Usual care for COPD includes oxygen therapy, steroid therapy, chest radiography, nebulized bronchodilators, and antimicrobial therapy.

INTERVENTIONS:
Behavioral: Get Palliative Care: four educational learning module videos — Organizational Sponsored public domain educational videos
  Arms: Get Palliative Care: four educational learning module videos

SUMMARY:
The goal of this pilot randomized controlled trial is to compare health literacy (HL) and quality of life (QOL) among older adults with chronic obstructive pulmonary disease (COPD) who completed a series of standardized palliative care (PC) educational video learning modules to usual care (US). The main question[s] it aims to answer are:

Between Groups:

* What effect does completing a series of standardized PC education video learning modules have on HL among older adults with COPD treated in the emergency department (ED) compared to usual care?
* What effect does completing a series of standardized PC education video learning modules have on QOL among older adults with COPD treated in the ED compared to usual care?

Within Groups:

* What is the change from baseline to study completion for older adults with COPD who receive the educational intervention series of PC learning modules on HL?
* What is the change from baseline to study completion for older adults with COPD who receive the educational intervention series of PC learning modules on QOL?
* What is the change from baseline to study completion for older adults with COPD who receive UC on HL?
* What is the change from baseline to study completion for older adults with COPD who receive UC on QOL?

All participants will complete a baseline and study completion health literacy questionnaire (HLQ) and Medical Outcomes Study: Short Form 36 survey. The treatment group will view one standardized learning module per week for four weeks provided by Get Palliative Care and log their weekly completion in REDCap. The control group will receive usual COPD care. Researchers will compare the treatment group receiving weekly palliative care education to usual care to see if HL and QOL change.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to conduct a pilot randomized controlled trial (RCT) to compare health literacy (HL) and quality of life (QOL) among older adults with chronic obstructive pulmonary disease (COPD) who completed a series of standardized palliative care (PC) educational video learning modules to usual care. Problem: Older adults aged 65 years and older with COPD are living longer, reported one in four have low HL, overall poorer health, and often seek emergency department (ED) care for the relief of symptoms impacting their QOL. Significance: The incidence of aging, the risk for chronic disease development like COPD with unpredictable disease trajectories, increased end-of-life healthcare costs, and limited HL have resulted in poor QOL. Limited research has been conducted on HL related to PC in the ED. Innovation: The pilot RCT will be a unique contribution to critical care nursing research by demonstrating the importance HL has on PC while improving overall QOL for older adult COPD patients seeking care in the ED. A 2030 Healthy People initiative is to decrease ED visits for COPD. Theory: The Expanded Chronic Care Model incorporates PC constructs focusing on older adults at risk for poor health outcomes while adding emphasis on digital constructs and educational training programs. Design: The study design is pilot RCT comparing QOL and HL among older adults with COPD treated in the ED who complete a series of standardized PC educational learning modules compared to usual care (UC). Setting: The study will be conducted at Missouri Baptist Medical Center, a community-based geriatric-designated ED in Saint Louis, Missouri. Sample: A convenience sample of older adults aged 65 or older with a diagnosis of COPD who seek care in the ED is the target population. This is a pilot study and, therefore, will have no statistical power with the overall goal of enrolling 30 participants. Intervention: All consenting participants will complete a baseline and study completion HL questionnaire (HLQ) and QOL survey. The treatment group will view one standardized learning module per week for four weeks provided by Get Palliative Care and log their weekly completion in REDCap. The control group will receive usual COPD care. Procedure: Informed consent will be obtained from participants who meet inclusion criteria and volunteer to participate in the study. Recruitment will take place for 30 days, and the study duration will be 30 days from the time of enrollment. A 1:1 randomization will be used to assign participants to the intervention or control group. Instrument: The Medical Outcomes Study Short Form-36 QOL survey and HLQ will measure the outcome variables at baseline and study completion. Analysis Plan: Demographic data using descriptive statistics will be calculated. Trends of the mean scores from baseline to study completion among groups and between groups will be conducted. REDCap will securely store all study-related data.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* COPD diagnosis
* English speaking
* Access to technology and Internet/online services

Exclusion Criteria:

* Enrolled in hospice care
* Cancer diagnosis stage IV or greater

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Health Literacy Questionaire | Baseline and immediately after the intervention, through study completion up to 12 weeks
  The HLQ has been validated for sample participants 65 years and older. The prose of the tool includes numeracy and comprehension. There are nine scales of multidimensional constructs of health and each scale is reliable and generates key information about an individual's perceived health literacy abilities, and their experiences. It was designed to be sensitive to change, identifying small differences between populations, and changes over time. The first five scales comprise items that ask the respondents to indicate their level of agreement on one of four response options (strongly disagree to strongly agree). The remaining scales (6-9) represent scales of self-reported capability and items within these scales are scored on one of five response options (cannot do; very difficult; quite difficult; quite easy; very easy).
Medical Outcomes Study-Short Form 36 | Baseline and immediately after the intervention, through study completion up to 12 weeks
  The Medical Outcomes Study Short Form-36 (SF-36) survey measures eight health concepts including physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, energy/fatigue levels, emotional well-being, social functioning, and vitality to measure quality of life. The SF-36 survey uses a 5-point Likert scale ranging from one which is equivalent to poorer (or poor) health to five which is equivalent to excellent health. Lower scores represent poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Lasiter, PhD, Study Chair — University of Missouri, Kansas City
Locations (1):
- Missouri Baptist Medical Center, St Louis, Missouri, United States